CLINICAL TRIAL: NCT02259881
Title: Investigation of the Effect of 0.9, 2.25 or 4.5 mg of BIBT 986 Over 1 Hour, Followed by 0.2, 0.5 or 1.0 mg/Hour of BIBT 986 for 7 Hours Given as IV Infusion on Tissue Factor Triggered Coagulation in a Randomised, Placebo Controlled, Dose Escalation Design in Healthy Male Volunteers
Brief Title: Effect of BIBT 986 Followed by BIBT 986 Given as IV Infusion on Tissue Factor Triggered Coagulation in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1192.11
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Lipopolysaccharides

ARMS (4):
- Low dose of BIBT 986 CL (Experimental)
  Interventions: Drug: Low dose of BIBT 986 CL, per i.v. infusion; Drug: Lipopolysaccharide (LPS), single i.v. bolus
- Medium dose of BIBT 986 CL (Experimental)
  Interventions: Drug: Medium dose of BIBT 986 CL, per i.v. infusion; Drug: Lipopolysaccharide (LPS), single i.v. bolus
- High dose of BIBT 986 CL (Experimental)
  Interventions: Drug: High dose of BIBT 986 CL, per i.v. infusion; Drug: Lipopolysaccharide (LPS), single i.v. bolus
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Lipopolysaccharide (LPS), single i.v. bolus

INTERVENTIONS:
Drug: Low dose of BIBT 986 CL, per i.v. infusion
  Arms: Low dose of BIBT 986 CL
Drug: Medium dose of BIBT 986 CL, per i.v. infusion
  Arms: Medium dose of BIBT 986 CL
Drug: High dose of BIBT 986 CL, per i.v. infusion
  Arms: High dose of BIBT 986 CL
Drug: Placebo
  Arms: Placebo
Drug: Lipopolysaccharide (LPS), single i.v. bolus — Endotoxin derived from E. coli bacteria, used for activation of coagulation

SUMMARY:
To compare with placebo the anticoagulant activity of three dosages of BIBT 986 on parameters of coagulation, platelet activation and inflammation in a model of tissue factor triggered activation of the coagulation system; to examine the safety of BIBT 986 in this setting

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by the screening procedure
* Signed written informed consent form in accordance with good clinical practice (GCP) and local legislation was available
* Age ≥ 18 and ≤ 40 years
* Body mass index: BMI ≥ 18 and ≤ 29.9 kg/m2
* Normal findings in medical history and physical examination unless the investigator considered an abnormality to be clinically irrelevant
* Normal laboratory parameters unless the investigator considered an abnormality to be clinically irrelevant

Exclusion Criteria:

* Any finding in the medical examination (including blood pressure, pulse rate, ECG, and laboratory parameters) deviating from normal and of clinical relevance
* History of or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, autoimmune, hormonal disorders, diseases of the central nervous system (such as epilepsy), or psychiatric disorders
* Symptoms of a clinically relevant illness in the 3 weeks before the first trial day
* History of orthostatic hypotension, fainting spells, and blackouts
* Chronic or relevant acute infections
* History of allergy / hypersensitivity (including drug allergy) which was deemed relevant to the trial as judged by the investigator
* History of

  * any bleeding disorder including prolonged or habitual bleeding
  * any familial bleeding disorder
  * other haematological disease
  * cerebral bleeding (e.g. after a car accident)
  * commotio cerebri
* Hereditary deficiency of protein C or S, or a mutation of factor V (Leiden), or any other known abnormality affecting coagulation, fibrinolysis, or platelet function
* Platelet count < 150000/μL
* Any ECG value outside of the reference range of clinical relevance (QRS interval > 110 ms or QTcB (QT interval Bazett correction) > 450 ms will be an obligatory exclusion criterion)
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs that might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Participation in an LPS trial within the last six weeks
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Concurrent or history of drug, alcohol, tobacco or coffee / tea / cola abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Seropositivity for hepatitis B surface antigen (HBs-Ag), hepatitis C virus (HCV), HIV 1, or HIV 2 antibodies
* Weight over 95 kg

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2002-12; Primary Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Change in activated partial thromboplastin time (aPTT) | up to 48 hours after start of treatment
Change in international normalized ratio (INR) | up to 48 hours after start of treatment
Change in thrombin time (TT) | up to 48 hours after start of treatment
Change in ecarin clotting time (ECT) | up to 48 hours after start of treatment
Change in prothrombin fragment (F1+2) | up to 48 hours after start of treatment
Change in D-dimer | up to 48 hours after start of treatment
Change in thrombin anti-thrombin complexes (TAT) | up to 48 hours after start of treatment
Change in protein C activity | up to 48 hours after start of treatment
Change in antithrombin | up to 48 hours after start of treatment
Change in thrombomodulin | up to 48 hours after start of treatment
Change in tissue factor messenger RNA (mRNA) | up to 48 hours after start of treatment
Change in platelet count | up to 48 hours after start of treatment
Change in plasmin antiplasmin complexes (PAP) | Pre-dose, up to day 14 after start of treatment
Change in soluble P-selectin | up to 48 hours after start of treatment
Change in tumor necrosis factor alpha (TNF alpha) | up to 48 hours after start of treatment
Change in interleukin-6 (IL-6) | up to 48 hours after start of treatment
Change in primary haemostasis measured by closure times | up to 48 hours after start of treatment
Number of subjects with clinically relevant changes in vital signs | up to 14 days after start of treatment
  blood pressure, pulse rate, body temperature
Number of subjects with clinically relevant changes in laboratory parameters | up to 14 days after start of treatment
Number of subjects with adverse events | up to 14 days after start of treatment
Number of subjects with clinically relevant changes in ECG | up to 14 days after start of treatment
Change in thrombus precursor protein | up to 48 hours after start of treatment
Change in soluble E-selectin | up to 48 hours after start of treatment

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | up to 48 hours after start of treatment
Maximum concentration in plasma at the end of the infusion (Cgh) | up to 48 hours after start of treatment
Apparent terminal half-life of BIBT 986 in plasma (t1/2) | up to 48 hours after start of treatment
Mean residence time of BIBT 986 in the body after intravenous bolus administration (MRT) | up to 48 hours after start of treatment
Volume of distribution of BIBT 986 in plasma at steady state (Vss) | up to 48 hours after start of treatment
Apparent volume of distribution of BIBT 986 during the terminal phase after intravenous infusion (Vz) | up to 48 hours after start of treatment